CLINICAL TRIAL: NCT03733275
Title: Efficacy of Preoperative Lidocaine Spray and Local Aensthetics-soaked Nasal Packings on Postoperative Pain After Nasal Closed Reduction
Brief Title: Efficacy of L/A Spray andL/A-soaked Nasal Packings on Postoperative Pain After Nasal Closed Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: yemoon
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Nasal Fracture
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- local anesthetic group (Experimental): local aensthetic group receive preopetaive lidocaine spray and lidocaine-bupivacine mixture-soaked nasal pacing after nasal reduction surgery
  Interventions: Drug: Lidocaine
- control group (Placebo Comparator): control group receive preoperative normal saline spray and normal saline-soaked nasal packing after nasal reduction surgery
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — for experimental arm, lidocaine spray and lidocaine bupivacine mixture-soaked nasal packing vs. for placebo arm, normal saline spray and packing
  Other Names: bupivacaine

SUMMARY:
This study is perfored to investigate the efficacy of preoperative lidocaine spray and lidocaine-bupivacaine mixture-soaked nasal packing for acute postoperative pain after nasal closed reduction surgery.

DETAILED DESCRIPTION:
To investigate the treatment of postoperative pain after nasal closed reduction surgery, we plan to investigate the effect of preoperative lidocaine spray and lidocaine-bupivacaine mixture-soaked nasal packing for the patinets undergoing nasal closed reduction under general aensthesia, compaing to the control group (normal saline spray and normal saline-soaked nasal packing).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to receive nasal reduction surgery under general aensthesia

Exclusion Criteria:

* concomitant disorders (eg. facial bone fractures) concomitant surgery (eg. septoplasty)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
postoperative pain in recovery room | immediately after surgery
  Using VAS, postoperative pain is measured.

SECONDARY OUTCOMES:
rescue analgesics in recovery room | 1 hr after surgery
  Fentanyl iv injection for pain control is checked.

CONTACTS AND LOCATIONS:
Overall Officials: Young Eun Moon, MD, Principal Investigator — Associate Professor
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided